CLINICAL TRIAL: NCT02640027
Title: Telemedicine in Supracondylar Humerus Fractures
Brief Title: The Use of Telemedicine Tool in Supracondylar Humerus Fractures in Children
Acronym: T-SCHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Mauricio Silva, Clinical Professor of Orthopaedics, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2015-12-16; First posted 2015-12-28 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Humeral Fractures
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment in the Clinic Only (No Intervention): Patients in Group A will receive their follow-up care entirely at the investigators institution
- Treatment in the Clinic and at Home (Experimental): Cast removal at home using a telemedicine tool
  Interventions: Procedure: Cast removal at home using a telemedicine tool

INTERVENTIONS:
Procedure: Cast removal at home using a telemedicine tool — Instead of receiving follow up treatment in a clinical setting, patients randomized to the arm of the study requiring telemedicine will receive some of their follow up care at home.
  Arms: Treatment in the Clinic and at Home

SUMMARY:
Fractures of the supracondylar region of the humerus are among the most common pediatric injuries requiring the attention of an orthopaedic surgeon. Children with non-displaced fractures (Type I), as well as those with history of elbow trauma, have been traditionally managed with non-surgical immobilization. Recently published clinical guidelines support such practice, based on the result of two prospective studies in which either collar and cuff or posterior splint immobilization were used. When compared to collar and cuff immobilization, posterior splints resulted in better pain relief within the first two weeks of injury; however, critical outcomes, including the incidence of cubitus varus, hyperextension, and loss of reduction, were not reported.

While posterior splints appear to be an attractive option for the treatment of non-displaced pediatric elbow fractures, a recent retrospective analysis on the use of posterior splints for the treatment of such injuries reported a small proportion of fractures demonstrating displacement. The potential for non-compliance with the use of removable devices, especially in the older pediatric population, is also a concern.

The use of a removable immobilization that can reliably maintain fracture alignment, minimize the risk of non-compliance, and result in similar outcomes as those obtained with regular casting could be advantageous: It appears that such immobilization could be removed easily and safely at home, potentially resulting in a lower number of patient visits, decreased health-care costs, and higher patient/parent satisfaction.

Telemedicine, defined as the use of telecommunication and information technologies in order to provide clinical health care at a distance, has been seldom used in the field of pediatric orthopaedics. Commonly mentioned attributes of telemedicine include improved access to healthcare providers, cost containment and increased healthcare efficiency, quality care improvements related to patient satisfaction, and potential reduction in travel time for patients and families.

The purpose of this randomized, controlled, prospective study is to assess telemedicine as a tool for the treatment follow-up of non-displaced SCHF fractures in children. Investigators hypothesize that using telemedicine will result in comparable clinical outcomes as those obtained in patients treated in a clinical facility, with increased patient satisfaction and decreased healthcare costs.

DETAILED DESCRIPTION:
The investigators will conduct an IRB approved, single-center, randomized, open label trial, in which children who present to the investigators institution with a non-displaced (Type 1) SCHF or an occult elbow injury (as determined by the presence of a posterior fat pad sign) will receive a long-arm soft, fiberglass cast (reinforced with a posterior slab) (3MTD "ScotchcastTM" Soft Cast Casting Tape) with the elbow flexed to 90-100 degrees and with forearm in neutral rotation and will be randomized to one of two groups: Patients in Group A will receive their follow-up care entirely at the investigators institution, while patients in Group B will receive some of the follow-up care using a telemedicine tool. Written informed consent will be obtained from the parents of each patient. For patients between the ages of seven and ten years, child assents will also be obtained.

Randomization will be accomplished by using sealed envelopes, sequentially numbered on the outside, in which a random sequence of A or B will be concealed. Sample size estimation was based on the outcome variable of percent average total satisfaction score. The investigators own previous studies at OIC presented a standard deviation of the satisfaction score of 15%. Clinically significant differences in satisfaction scores were on the order of 10 to 15%. In the present study, 25 patients in each group will be included, for a total of 50 patients. With this sample size, the investigators will be able to detect differences of 12% in satisfaction score with alpha of 0.05 and 80% power.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 2 and 10 years (open physis), who present within seven days of sustaining a closed, non-displaced, type I supracondylar humeral fracture or a closed, acute elbow injury in whom a fracture is not seen but a positive posterior fat pad sign is identified will be considered for inclusion in the present study. In order to be included, the patient's family must have access to an electronic device with a camera (desktop computer, laptop, tablet or cell phone) with internet connectivity, and be willing to download and use a free application for live videoconferencing (WebEx, Cisco Systems). WebEx is a HIPPA compliant videoconferencing system that includes audio and visual components.

Exclusion Criteria:

* Patients younger than 2 or older than 10 years of age will be excluded, as well as those with a displaced or open elbow fracture, any associated generalized condition that affects the elbow range of motion, history of a previous injury or surgery to the elbows, a neurovascular abnormalities or suspicion of a compartment syndrome or a pathological fracture.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Fracture displacement as measured by Baumann Angle | At 8 week follow up visit
  Fracture displacement will be assessed by comparing the initial values of the Baumann angle of the elbow, taken at the 1 week follow up visit, with those obtained during the 8th week follow-up appointment.
Fracture angulation as measured by Shaft Condylar Angle | At 8 week follow up visit
  Fracture angulation will be assessed by comparing the initial values of the shaft-condylar angle of the elbow, taken at the 1 week follow up appointment, and the position of the anterior humeral line with respect to the capitellum, with those obtained during the 8th week follow-up appointment.

SECONDARY OUTCOMES:
Recovery of Range of Motion Using a 6" E-Z Read Jamar® Goniometer | 8 Weeks after injury
  The recovery of ROM will be assessed at the 8th week follow-up by comparing the range of motion of the affected elbow with that of the normal, contralateral elbow. The range of motion of the elbow will be measured with the use of a small goniometer calibrated in 1° increments, using standard techniques. All ROM measurements will be performed by a single observer using the same goniometer.
Elbow Pain Using the Revised Faces Pain Scale | Weeks 4 and 8 after injury
  Elbow pain will be measured at weeks 4 and 8 with the use of the Faces Pain Scale. This is a validated, highly reliable scale, commonly used in the pediatric population. Hicks CL, von Baeyer CL, Spafford PA, et al. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001;93:173-183.